CLINICAL TRIAL: NCT06994689
Title: Clinimetric Properties Assessment of Quadriceps Muscle Mass and Stiffness Using Perimetry and ShearWave Elastography in Patients With COPD : a Prospective Observational Study
Brief Title: Clinimetric Properties of Muscle Mass and Stiffness Measurements of the Quadriceps in Patients With COPD
Acronym: Metriquad
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier du Havre (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00297-36
Record Dates: First submitted 2025-03-27; First posted 2025-05-29 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COPD; Quadriceps Muscle Atrophy
Keywords: Clinimetric properties; Muscle mass; Muscle strength
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Visual Field Tests; Electric Impedance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Perimetry and ShearWave measurement of the quadriceps muscle before and after a pulmonary rehabilitation (PR) programme — Patients will undergo a pulmonary rehabilitation (PR) programme.
  On day 1, perimetry and ShearWave measurements of the quadriceps muscle will be provided. Supplementary assessments of quadriceps thickness, quadriceps strength with a handheld dynamometry, lean body mass (bioelectrical impedance), constant work-rate endurance test and HAD questionnaire will also be provided on day 1.
  The same measurements and questionnaire will be provided on the last day of the patient in the PR programme.
  Other Names: Functional exercice capacity; Quality of life; Bioelectrical impedance; Quadriceps thickness; Quadriceps strength : maximal voluntary contraction

SUMMARY:
A large amount of patients with COPD suffer from muscle dysfunction characterized by losses of muscle mass and strength. Studies have shown an association between a loss of quadriceps muscle mass and premature death.

This study aims to investigate the clinimetric properties of a simple quadriceps perimetry and ShearWave elastography to improve the monitoring of skeletal muscle function in patients with COPD.

DETAILED DESCRIPTION:
Muscle dysfunction in COPD is characterized by reduced skeletal muscle mass and strength, particularly in the lower limbs. These systemic consequences of COPD play a key role in the course of these patients, through their impact on functional status, quality of life and increased mortality. Early detection and monitoring of muscular status in these patients could help improve management and limit the consequences of the disease.

Numerous studies show that variation in quadriceps mass has a significant relationship with premature mortality in this disease. The use of an indirect but simple and affordable measure: perimetric tape-measurement of thigh circumference, could help monitor quadriceps muscle mass in these patients on a regular and cost-effective basis. However, the clinimetric properties (validity, reliability, response to treatment) of this measurement need to be assessed to clarify its relevance.

On the other hand, ShearWave ® elastography (SWE) is a new method of measuring quadriceps stiffness. This measurement could provide additional information on muscle quality compared with conventional measures of strength or muscle trophicity. The potential added value of SWE ® for COPD patients has not yet been investigated. This tool would provide more precise indications of the state of the quadriceps, with the aim of improving the management of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients
* Adults (>18 years old)
* Patients starting a pulmonary rehabilitation (PR) programme

Exclusion Criteria:

* Patients included in other research protocol
* Minors or under guardianship
* Pregnancy
* Patients with lower limb amputation or history of neuromuscular disease
* Cardiovascular contradications for PR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients completing a PR programme for 5 weeks
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Perimetry of the quadriceps | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  Thigh circumference measured by a tape
Quadriceps stiffness | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  ShearWave elastography of the quadriceps muscle

SECONDARY OUTCOMES:
Lean body mass | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  measured by bioelectrical impedance
Functional exercise capacity | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  measured as the endurance time during a constant load endurance test using a cycloergometer or a treadmill
Health-Related Quality of Life | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  measured by quality of life questionnaire (hospital anxiety and depression scale (HAD))
Quadriceps thickness | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  measured by ultrasonography
Quadriceps strength | At day 1 and after 5 weeks (at the end of the 5 weeks pulmonary rehabilitation program)
  measure of maximal voluntary contraction with handheld dynamometry

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier du Havre, Le Havre, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning after publication and ending 60 months following article publication.
Access Criteria: For individual participant data meta-analysis. Proposals should be directed to yann.combret@gmail.com. To gain access, data requestors will need to sign a data access agreement.